CLINICAL TRIAL: NCT02388776
Title: Use of Rotational Thromboelastometry (ROTEM) to Characterize Coagulation Abnormalities in Burn Patients: A Prospective Pilot Study
Brief Title: Use of Rotational Thromboelastometry (ROTEM) to Characterize Coagulation Abnormalities in Burn Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subject recruitment unable to be completed due to study feasibility issues.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1404014977
Record Dates: First submitted 2015-02-02; First posted 2015-03-17 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Burn
Keywords: ROTEM; Fibrinogen
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ROTEM (Experimental): Clinical burn ICU Inpatients receiving blood draws for ROTEM analysis and fibrinogen levels.
  Interventions: Device: ROTEM

INTERVENTIONS:
Device: ROTEM — A blood sample and reagents are placed into a small cup. A pin suspended from a wire is immersed into the sample. The pin rotates back and forth at a fixed angle. The movement of the pin is optically monitored and converted into a real time measurement that is represented graphically. Prior to clot formation, pin rotation is unhindered and is graphically represented as a straight line. As the subject's blood sample starts to clot, strands of clot form between the pin and the cup wall, restricting the movement of the pin depending on the strength of the clot. Graphically, this is represented as a symmetrical widening of the curve.
  Other Names: ROTEM delta

SUMMARY:
This is an interventional pilot study of 40 burn inpatients. Specific aims of the proposed pilot study are to use bedside blood analysis with rotational thromboelastometry (ROTEM) in severe burn patients to provide preliminary information on the nature of coagulation abnormalities and compare subject ROTEM coagulation profiles within 24 hours of burn injury (day 1) and on days 2, 3, 5, 7, 14 and 21 after burn injury.

DETAILED DESCRIPTION:
Specific aims of this pilot study are to use bedside blood analysis with ROTEM in severe burn patients to provide preliminary information on the nature of coagulation abnormalities and to compare subject ROTEM coagulation profiles within 24 hours of burn injury (day 1) and on days 2, 3, 5, 7, 14 and 21 after burn injury. Investigators hypothesize that ROTEM analysis will detect a pattern of impaired coagulation in severely burned patients.

ROTEM analysis:

A blood sample and reagents are placed into a small cup. A pin suspended from a wire is immersed into the sample. The pin rotates back and forth at a fixed angle. The movement of the pin is optically monitored and converted into a real time measurement that is represented graphically. Prior to clot formation, pin rotation is unhindered and is graphically represented as a straight line. As the subject's blood sample starts to clot, strands of clot form between the pin and the cup wall, restricting the movement of the pin depending on the strength of the clot. Graphically, this is represented as a symmetrical widening of the curve. Blood will be obtained for ROTEM/ fibrinogen levels from each subject seven times during their hospital admission: once within 24 hours of burn injury (day 1), and on days 2, 3, 5, 7, 14 and 21. For each sample, 5.4 mL of whole blood will be collected into 2 citrated tubes (2.7 mL in each tube). For all subjects, both pediatric and adult, blood will be collected via an indwelling catheter (arterial or central line). One 2.7 ml tube will be used for ROTEM analysis. The amount of blood is in accordance with the acceptable limit of ROTEM analysis. ROTEM testing will be performed according to the manufacturer's instructions using test kit reagents. Members of the clinical research team who have been trained and certified to use the ROTEM device will perform the appropriate ROTEM tests. The second 2.7 mL citrated tube will be used to measure fibrinogen level, using the automated central laboratory device in hospital.

In this interventional study, the ROTEM data will be blinded to the treating Burn ICU physicians and will have no effect on standard perioperative and ICU treatment. The ROTEM machine will be located in a designated spot outside of the ICU, out of view of the treating clinicians. Thus, volume replacement, thrombosis prophylaxis, and other management (including blood product transfusions) will be performed according to existing protocols.

Demographic information will be de-identified, but will include demographics (age, sex) and each subject's medical and surgical history, burn injury type (thermal, chemical, electrical, inhalational, plus/minus additional injury - i.e. Trauma/TBI, etc) and percent Total Body Surface Area (TBSA) as diagrammed by the Burn ICU on admission, medications (specifically, form of venous thromboembolism prophylaxis as prescribed by ICU physicians during the study period), weight, vital signs, dates of surgical intervention (bedside escharotomies and OR procedures), dates and types of blood product administration, fluid balance per day, number of days intubated, number of ICU days, hospital LOS, mortality, and ISS. Laboratory values: (on days 1, 2, 3, 5, 7, 14, and 21) will include fibrinogen, PT, INR, aPTT, and CBC when available as standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients admitted to NYPH with 15% TBSA burn or greater.
2. Patients with vascular access catheters (arterial or central line) placed within 24 hours of burn injury
3. Males and females
4. Ages >3 years or >15 kg
5. Informed verbal consent obtained from the patient or the patient's designated health care proxy (DHCP). In the case of minors, assent and informed verbal consent obtained from at least one parent or guardian.

Exclusion Criteria:

1. Known pre-existing hemostatic abnormalities
2. Ages < 3 years or weight < 15 kg
3. Intake of anticoagulants or antiplatelet aggregation inhibitors prior to burn
4. Pregnant patients
5. Patients with delayed presentation (greater than 24 hours after burn injury)
6. Inclusion in another clinical research study
7. Refusal or inability of patient or patient's DHCP to consent in English.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lennon, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ROTEM
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | ROTEM
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Coagulation Parameters
Description: To compare ROTEM coagulation parameters involving fibrin contribution to clot formation (FIBTEM) between patients on admission/enrollment (day 1), and on days 2, 3, 5, 7, 14 and 21 after burn injury to see if expected hypercoagulability shows evidence of resolution.
Time Frame: 21 days
Population: Data not collected for two subjects for all time points for primary outcome due to subject being discharged from hospital and subject death.
Groups:
- Active Arm: Clinical burn ICU Inpatients receiving blood draws for ROTEM analysis and fibrinogen levels.
  ROTEM: A blood sample and reagents are placed into a small cup. A pin suspended from a wire is immersed into the sample. The pin rotates back and forth at a fixed angle. The movement of the pin is optically monitored and converted into a real time measurement that is represented graphically. Prior to clot formation, pin rotation is unhindered and is graphically represented as a straight line. As the subject's blood sample starts to clot, strands of clot form between the pin and the cup wall, restricting the movement of the pin depending on the strength of the clot. Graphically, this is represented as a symmetrical widening of the curve.
Arm/Group | Active Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Predictive Value of ROTEM Data
Description: To assess whether ROTEM abnormalities correlate with allogenic blood product administration by blinded ICU physicians
Time Frame: 21 days
Population: Only two subjects enrolled, one withdrawn early due to death and the second lost to follow up prior to the completion of the final ROTEM testing.
Arm/Group | ROTEM
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a five month period.
Description: Serious adverse events were defined as Grade 3-5 events, as defined by the NIH. All other adverse events were events defined as Grade 1-2.
Arm/Group | Active Arm
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Arm (N=2)
Respiratory failure; grade 4 (Respiratory, thoracic and mediastinal disorders) | 1
Contusion/pneumonia; grade 3 (Respiratory, thoracic and mediastinal disorders) | 1
SIRS; grade 3 (Immune system disorders) | 1
Anuria; grade 4 (Renal and urinary disorders) | 1
Metabolic acidosis; grade 4 (Metabolism and nutrition disorders) | 1
Hemachromaturia (Metabolism and nutrition disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Massive anasarca (Skin and subcutaneous tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Arm (N=2)
Protein calorie malnutrition (Metabolism and nutrition disorders) | 1
Abnormal lab value/low hemoglobin (Blood and lymphatic system disorders) | 1
Abnormal lab value/low hematocrit (Blood and lymphatic system disorders) | 1
Abnormal lab value/high INR (Blood and lymphatic system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Cellulitis (Infections and infestations) | 1
Hypermetabolism (Metabolism and nutrition disorders) | 1
Abnormal lab value/hemoglobin dropped from 8.2 to 7 (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 1
MSSA and Klebsiella (Infections and infestations) | 1
Abnormal lab value/high sodium and uptrending creatinine (Blood and lymphatic system disorders) | 1
Thermal keratopathy, right eye (Eye disorders) | 1
Bilateral upper and lower eyelid swelling (Eye disorders) | 1
Cardiac ischemia (Cardiac disorders) | 1
Red blood per rectum (Gastrointestinal disorders) | 1
Pleural fluid (Respiratory, thoracic and mediastinal disorders) | 1
Hypothermia (General disorders) | 1
Leukopenia (Immune system disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Small numbers of subjects due to the critical condition of subject population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes